CLINICAL TRIAL: NCT04088279
Title: Novel Quantitative Magnetic Resonance Imaging (MRI) Measures in the Assessment and Follow-up of Patients With Pulmonary Hypertension (PH)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 246688
Record Dates: First submitted 2019-07-31; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Hypertension
Keywords: MRI; oxygen enhanced; fourier decomposition
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI — Oxygen enhanced and fourier decomposition MRI

SUMMARY:
A prospective study of the use of two novel MRI techniques (oxygen-enhanced and fourier decomposition MRI) in the initial diagnosis and follow-up of patients with Pulmonary Hypertension. The investigators believe these techniques may present a novel set of imaging biomarkers that may be used for risk stratification, prediction of treatment response and longitudinal disease monitoring. The reserach MRI is in addition to standard of care and will not affect treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Pulmonary Hypertension.
* Age 18 and over.

Exclusion Criteria:

* Standard contra-indications to MRI (as per NHS MRI safety questionnaire).
* Not medically fit for transfer to MRI.
* Patient judged inappropriate for involvement in study by clinical team e.g. secondary to emotional burden of recent diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Delta pO2 max (mmHg) | Baseline and 3-6 months
Wash in and wash out time constants (min) | Baseline and 3-6months
Signal Intensity Change (%) | Baseline and 3-6months
Fractions (% area of lung imaged) | Baseline and 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Simon Padley, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No